CLINICAL TRIAL: NCT03551743
Title: A Randomized, Double-Blind, Vehicle-Controlled Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered PRT064445 After Dosing to Steady State With One of Four Direct/Indirect fXa Inhibitors in Healthy Volunteers
Brief Title: Phase 2 Healthy Volunteer Study to Evaluate the Ability of PRT064445 to Reverse the Effects of Several Blood Thinner Drugs on Laboratory Tests (Module 4 of 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-502 Module 4
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PRT064445; edoxaban

STUDY DESIGN:
Intervention Model Description: This study has four modules with a total of 21 cohorts, each module was reported and submitted separately.
  Module 1, NCT01758432 (54 subjects with 7 cohorts including placebo); Module 2, NCT03578146 (48 subjects with 6 cohorts including placebo); Module 3, NCT03551730 (27 subjects with 4 cohorts including placebo); Module 4, NCT03551743 (28 subjects with 4 cohorts including placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Module 4 (600 mg bolus) (Experimental): 600 mg PRT064445 given as a single IV bolus
  Interventions: Combination Product: PRT064445/Edoxaban; Combination Product: Placebo/Edoxaban
- Module 4 (800 mg bolus + 480 mg infusion) 8mg/min (Experimental): 1280 mg PRT064445: 800 mg IV at ~30 mg/min, followed by a continuous infusion of 480 mg (4 mg /min over 60 minutes)
  Interventions: Combination Product: PRT064445/Edoxaban; Combination Product: Placebo/Edoxaban
- Module 4 (800 mg bolus) (Experimental): 800 mg PRT064445 as a single IV bolus
  Interventions: Combination Product: PRT064445/Edoxaban; Combination Product: Placebo/Edoxaban
- Module 4 Placebo (Placebo Comparator): Placebo administered intravenously (IV) as a bolus or a bolus followed by continuous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: PRT064445/Edoxaban
  Other Names: Andexanet
  Arms: Module 4 (600 mg bolus); Module 4 (800 mg bolus + 480 mg infusion) 8mg/min; Module 4 (800 mg bolus)
Combination Product: Placebo/Edoxaban
  Arms: Module 4 (600 mg bolus); Module 4 (800 mg bolus + 480 mg infusion) 8mg/min; Module 4 (800 mg bolus)
Drug: Placebo
  Arms: Module 4 Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of PRT064445 to reverse the effects of several blood thinner drugs on laboratory tests. The study also is evaluating the blood levels of PRT064445 given at different doses.

DETAILED DESCRIPTION:
A randomized, double-blind, vehicle-controlled study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of intravenously administered PRT064445 after dosing to steady state with one of four direct/indirect factor Xa (fXa) inhibitors in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 45 years old

Exclusion Criteria:

* History (including family history) or symptoms of, or risk factors for bleeding
* History (including family history) of or risk factors for a hypercoagulable or thrombotic condition
* Absolute/relative contraindication to anticoagulation or treatment with specific anticoagulants
* History of major surgery, severe trauma or bone fracture within 3 months prior to dosing; or planned surgery within 1 month after dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

REFERENCES:
- [Derived] Lu G, Conley PB, Leeds JM, Karbarz MJ, Levy GG, Mathur VS, Castillo J, Crowther M, Curnutte JT. A phase 2 PK/PD study of andexanet alfa for reversal of rivaroxaban and edoxaban anticoagulation in healthy volunteers. Blood Adv. 2020 Feb 25;4(4):728-739. doi: 10.1182/bloodadvances.2019000885. PMID 32092140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative site in the US between March 2014 through August 2015
Pre-assignment Details: 28 subjects were enrolled in Module 4. Edoxaban was administered 60 mg orally once daily for 6 days in an open label fashion. Andexanet/placebo was administered intravenously (IV) on Day 6 such that they ended at 3 hours (Cohorts 1 and 2) or 5 hours (Cohort 3) after the last dose of edoxaban.
Groups:
- Module 4 (600mg): 600 mg andexanet IV bolus administered over ~20 minutes (~30 mg/min)
- Module 4 (800 mg Bolus + 480 mg Infusion): 800 mg andexanet IV bolus over ~27 minutes (~30 mg/min) followed immediately by a continuous infusion of 480 mg (8 mg/min over 60 min) [total 1280 mg]
- Module 4 (800 mg): 800 mg andexanet IV bolus administered over ~27 minutes (~30 mg/min)
Period: Overall Study
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Started | 10 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 28 subjects were enrolled in Module 4 and 26 subjects completed the study follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg) | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (8.35) | 38.8 (8.61) | 31.3 (8.82) | 35.5 (8.55) | 33.4 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 8
  Male | 8 | 4 | 5 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent Change From Baseline in Anti-fXa Activity at 2 Mins Following Andexanet/Placebo Administration
Description: Anti-fXa activity was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Anti-fXa activity was measured using a commercial kit (Coamatic Heparin-82 33 9363, DiaPharma)
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 26 subjects who received andexanet or placebo were included in the pharmacodynamics (PD) analysis
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
Percent change in anti-fXa activity | -27.64 (13.091) | -51.71 (15.95) | -72.60 (8.35) | -82.04 (6.66)
Statistical Analysis 1: Comparison: Module 4 Placebo vs Module 4 (600mg); Test type: Superiority; p = 0.0344, ANCOVA; Least Squares Means (Difference) = -65.02
Statistical Analysis 2: Comparison: Module 4 Placebo vs Module 4 (800 mg Bolus + 480 mg Infusion); Test type: Superiority; p = 0.0014, ANCOVA; Least Squares Means (Difference) = -92.38
Statistical Analysis 3: Comparison: Module 4 Placebo vs Module 4 (800 mg); Test type: Superiority; p = 0.0002, ANCOVA; Least Squares Means (Difference) = -46.26

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Thrombin Generation at 2 Mins Following Andexanet/Placebo Administration
Description: Thrombin generation was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Thrombin generation was measured using a TF-initiated thrombin generation assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 26 subjects who received andexanet or placebo were included in the PD analysis
Measure: Mean (Standard Deviation); unit: Percent change in thrombin generation
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
Percent change in thrombin generation | 18.09 (20.716) | 143.37 (31.742) | 252.92 (115.318) | 238.16 (82.287)
Statistical Analysis 1: Comparison: Module 4 Placebo vs Module 4 (600mg); Test type: Superiority; p = 0.0032, ANCOVA; Least Squares Means (Difference) = 88722.37
Statistical Analysis 2: Comparison: Module 4 Placebo vs Module 4 (800 mg Bolus + 480 mg Infusion); Test type: Superiority; p = 0.0003, ANCOVA; Least Squares Means (Difference) = 151500.3
Statistical Analysis 3: Comparison: Module 4 Placebo vs Module 4 (800 mg); Test type: Superiority; p = 0.0004, ANCOVA; Least Squares Means (Difference) = 198560.4

3. Secondary Outcome: Efficacy: Percent Change From Baseline in Unbound Edoxaban Plasma Concentration at 2 Mins Following Andexanet/Placebo Administration
Description: Unbound edoxaban concentrations was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Unbound plasma concentrations for edoxaban was determined by a rapid equilibrium dialysis method followed by Liquid chromatography- Mass Spectrometry.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 26 subjects who received edoxaban were included in the edoxaban pharmacokinetics (PK) analysis
Measure: Mean (Standard Deviation); unit: Percent change in unbound edoxaban conce
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
Percent change in unbound edoxaban conce | -17 (15) | -56 (7) | -66 (9) | -76 (13)
Statistical Analysis 1: Comparison: Module 4 Placebo vs Module 4 (600mg); Test type: Superiority; p = 0.1874, ANCOVA; Least Squares Means (Difference) = -76.05
Statistical Analysis 2: Comparison: Module 4 Placebo vs Module 4 (800 mg Bolus + 480 mg Infusion); Test type: Superiority; p = 0.386, ANCOVA; Least Squares Means (Difference) = -27.98
Statistical Analysis 3: Comparison: Module 4 Placebo vs Module 4 (800 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -49.99

4. Secondary Outcome: Andexanet Maximum Observed Plasma Concentration (Cmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Maximum observed plasma concentration was taken directly from the raw data.
Time Frame: Blood was collected at predose, 0.033, 0.2, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6.5, 7.5, 8.5 and 14.5 hours postdose.
Population: 18 subjects who received andexanet are included in the PK analysis for andexanet
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
ng/mL | NA (NA) — Andexanet was not administered (placebo group) | 111000 (20000) | 176000 (16600) | 235000 (106000)

5. Secondary Outcome: Andexanet Area Under the Drug Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf )
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. AUC0-inf was calculated using a non-compartmental approach
Time Frame: as for outcome 4
Population: 18 subjects who received andexanet are included in the PK analysis for andexanet
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Andexanet not administered (placebo group) | 129000 (26900) | 315000 (39600) | 241000 (77200)

6. Secondary Outcome: Andexanet Time of Maximum Observed Plasma Concentration (Tmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Tmax was taken directly from the raw data.
Time Frame: as for outcome 4
Population: 18 subjects who received andexanet are included in the PK analysis for andexanet
Measure: Median (Full Range); unit: hr
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
hr | NA [NA to NA] — Andexanet not administered (placebo group) | 0.38 [0.36 to 0.40] | 0.49 [0.49 to 0.74] | 0.50 [0.49 to 0.85]

7. Secondary Outcome: Andexanet Apparent Terminal Elimination Half-life (t1/2)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. t1/2 was determined by linear regression of the log concentration on the terminal portion of the plasma concentration-time curve.
Time Frame: as for outcome 4
Population: 18 subjects who received andexanet are included in the PK analysis for andexanet
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
hr | NA (NA) — Andexanet not administered (placebo group) | 8.21 (6.08) | 6.90 (1.57) | 8.06 (3.24)

8. Secondary Outcome: Andexanet Total Systemic Clearance (CL)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. CL was calculated using a non-compartmental approach.
Time Frame: as for outcome 4
Population: 18 subjects who received andexanet are included in the PK analysis for andexanet
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
L/hr | NA (NA) — Andexanet not administered (placebo group) | 4.80 (0.872) | NA (NA) — Not calculable, since parameter does not take into account the 60 minutes interval | 3.57 (0.995)

9. Secondary Outcome: Andexanet Total Volume of Distribution (Vss)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Vss was calculated using a non-compartmental approach.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Number analyzed (Participants) | 8 | 6 | 6 | 6
L | NA (NA) — Andexanet not administered (placebo group) | 6.16 (1.96) | NA (NA) — Not calculable, since parameter does not take into account the 60 minutes interval | 4.34 (1.61)

ADVERSE EVENTS:
Time Frame: ~7 weeks
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Groups:
- Module 4 Placebo: Placebo administered IV as a bolus or a bolus followed by continuous infusion.
Arm/Group | Module 4 Placebo | Module 4 (600mg) | Module 4 (800 mg Bolus + 480 mg Infusion) | Module 4 (800 mg)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 5/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Module 4 Placebo (N=8) | Module 4 (600mg) (N=6) | Module 4 (800 mg Bolus + 480 mg Infusion) (N=6) | Module 4 (800 mg) (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site hematoma (General disorders) | 0 | 0 | 1 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Conducted in healthy volunteers at Clinical Research Organization.